CLINICAL TRIAL: NCT02398682
Title: Acute Kidney Outreach to Reduce Deterioration and Death (AKORDD) - A Pilot Study to Look at Enhancing Patient Care, Improving Patient Outcomes and Reducing NHS Costs
Brief Title: Acute Kidney Outreach to Reduce Deterioration and Death (AKORDD)
Acronym: AKORDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heart of England NHS Trust (Other)
Collaborators: University of Birmingham (Other); University of Warwick (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PB-PG-1111-26038
Record Dates: First submitted 2015-03-20; First posted 2015-03-25 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Acute Kidney Injury
Keywords: electronic alerts; acute kidney injury; NHS; mortality
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- After study Intervention arm Heartlands (Experimental): The trial has 4 arms in a Before and After design:
  Arm 3. After/Heartlands area patients receiving the experimental intervention
  Patients who have AKI and are either inpatients in the Intervention hospital or living within the surrounding catchment area are eligible. The intervention will be in the form of a telephone call to the primary clinician or visit to the patient. The intervention will include:
  Rapid diagnosis of AKI cause; Rapid treatment of AKI cause; Stopping 'nephrotoxic' drugs; Early nephrology followup for stage 3 AKI survivors; and preventing recurrent AKI.
  Interventions: Other: Rapid diagnosis of AKI cause; Other: Rapid treatment of AKI cause; Other: Stopping 'nephrotoxic' drugs; Other: Early nephrology followup for stage 3 AKI; Other: Preventing recurrent AKI; Other: Good standard care
- After study Control arm Good Hope (Active Comparator): The trial has 4 arms in a Before and After design:
  Arm 4. After/Good Hope area patients observed whilst receiving active comparator
  Patients who have AKI, as shown by having an Alert for such, and are either inpatients in Good Hope Hospital or living within the surrounding catchment area. These patients will receive good standard care (active comparator), but none of the interventions listed for the Intervention group.
  Interventions: Other: Good standard care
- Before study Heartlands area (Active Comparator): The trial has 4 arms in a Before and After design:
  Arm 1. Before/Heartlands area patients observed whilst receiving active comparator
  Patients who have AKI, as shown by having an Alert for such, and are either inpatients in Heartlands Hospital or living within the surrounding catchment area. These patients will receive good standard care (active comparator), but none of the interventions listed for the Intervention group.
  Interventions: Other: Good standard care
- Before study Good Hope area (Active Comparator): The trial has 4 arms in a Before and After design:
  Arm 2. Before/Good Hope area patients observed whilst receiving active comparator
  Patients who have AKI, as shown by having an Alert for such, and are either inpatients in Good Hope Hospital or living within the surrounding catchment area. These patients will receive good standard care (active comparator), but none of the interventions listed for the Intervention group.
  Interventions: Other: Good standard care

INTERVENTIONS:
Other: Rapid diagnosis of AKI cause — The Outreach team will advise on an evidence-based package of care:
  1) Rapidly establish a credible diagnosis of the cause of AKI including:
  1. Improved assessment of volume status
  2. Standardised use of urine dipstick .
  3. Appropriate sepsis investigations.
  4. Urgent ultrasound with suspected obstruction.
  Arms: After study Intervention arm Heartlands
Other: Rapid treatment of AKI cause — Rapid, limited treatment of hypovolaemia, with avoidance of iatrogenic fluid overload, recently recognised as a significant cause of mortality in AKI. Rapid sepsis therapy. Urgent relief of urinary tract obstruction.
  Arms: After study Intervention arm Heartlands
Other: Stopping 'nephrotoxic' drugs — Cessation of all potentially nephrotoxic drugs.
  Other Names: Avoidance of iatrogenic causes of AKI
  Arms: After study Intervention arm Heartlands
Other: Early nephrology followup for stage 3 AKI — A rapid followup at discharge in an AKI clinic for survivors of stage 3 AKI, within 7 days of discharge for those in hospital, or within 7 days of the Alert for those not admitted to hospital.
  Arms: After study Intervention arm Heartlands
Other: Preventing recurrent AKI — Patients with AKI in the Intervention arm will receive information on preventing AKI during the study.
  Other Names: Patient information to reduce recurrent AKI
  Arms: After study Intervention arm Heartlands
Other: Good standard care — Good standard care will be provided for all patients in non Experimental arms; clinicians will continue to be able to rapidly refer patients for Nephrology advice or review; online guidance will be available for all clinicians and noted in the alerts for all cases of AKI.

SUMMARY:
The study pilots an outreach service for Acute kidney injury (AKI) patients, based on electronic alerts. Using the alerts we will contact the primary clinician caring for the patient with AKI in the Intervention group. The study has a control group of patients receiving good standard care, but without Outreach. The aim is to reduce morbidity and mortality in the syndrome, and also to reduce healthcare costs.

DETAILED DESCRIPTION:
Lay summary:

About one in six hospital inpatients suffer Acute Kidney Injury (AKI), also called acute renal failure. About a third of patients with AKI die. The large majority of patients with AKI are managed by doctors who are not kidney experts. Effective AKI advice and treatments are available but not currently integrated into routine care. A recent National review of the care of patients who died from AKI showed poor management of many patients. Early diagnosis of AKI can avoid complications, dialysis (which affects the quality of life of patients, and is costly) or death. AKI is diagnosed by a change in a blood test. We have developed computer software to diagnose AKI earlier. It sends a warning or 'Alert' about the test to our team of kidney experts. We will further develop the settings of the Alert system. It needs to send an Alert for the right patients. We will also study the best way to make clinicians pay attention to their patients who are developing AKI. When our expert Outreach team receive an Alert, they will call the doctor or nurse looking after the patient with AKI. We will advise on the best treatment for that patient, to reduce their risk of death, dialysis and other complications. We will do a pilot study in one large hospital, to further develop the system, and check it reduces the risk of death or complications from AKI. We will use this work to develop a larger trial of this new system of care for patients with AKI in different hospitals. This will convince the wider NHS of the need to change, and show how to prevent or reduce AKI. Ultimately we aim to improve patients' lives by reducing avoidable death and illness from AKI , and also save the NHS money.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with an Alert for AKI issued in accordance with the national algorithm for AKI alerts (NHS England)
* AKI stage 2 or 3 (this criterion is under review during the preparatory phase of the study)

Exclusion Criteria:

* patients already on dialysis for AKI at the time of alert
* patients with End stage renal disease
* patients <18 years of age
* patients with no evidence of AKI on review of the automated Alert
* patients dissenting from participation according to the Ethics application

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1865 (Actual)
Dates: Start 2014-10; Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Composite measure of participants not alive, need for dialysis, or progression of AKI stage | within 30 days
  Combined endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Mark Thomas, FRCP, Principal Investigator — Heart of England NHS Trust
Locations (1):
- Heart of England hospital NHS trust, Birmingham, Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Contact the Chief Investigator mark.thomas@heartofengland.nhs.uk

REFERENCES:
- [Derived] Abdelaziz TS, Lindenmeyer A, Baharani J, Mistry H, Sitch A, Temple RM, Perkins G, Thomas M. Acute Kidney Outreach to Reduce Deterioration and Death (AKORDD) trial: the protocol for a large pilot study. BMJ Open. 2016 Aug 19;6(8):e012253. doi: 10.1136/bmjopen-2016-012253. PMID 27543592